CLINICAL TRIAL: NCT00666835
Title: Randomized, Double-blind, Multicenter, Parallel-group, Equivalence Study to Evaluate the Efficacy and Safety of HX575 Hexal AG vs ERYPO® for the Treatment of Anemia in Hemodialysis Patients
Brief Title: Study to Evaluate the Efficacy and Safety of HX575 Hexal AG vs ERYPO® for the Treatment of Anemia in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-29-INJ-9
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Anemia
Keywords: Treatment of anemia in hemodialysis patients
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HX575 epoetin alfa Hexal AG (Experimental): Eligible patients were switched from the comparator ERYPO®, to epoetin alfa HX575 Hexal AG in ratio 2:1 to be intravenously treated with HX575 in pre-filled syringes for 24 weeks (solution for injection i.v.). The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL.
  Interventions: Drug: HX575 epoetin alfa Hexal AG
- ERYPO®, Janssen-Cilag (Active Comparator): Eligible patients were randomized and continued to be treated with ERYPO® Janssen-Cilag in pre-filled syringes intravenously (solution for injection i.v.) for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL.
  Interventions: Drug: ERYPO®, Janssen-Cilag

INTERVENTIONS:
Drug: HX575 epoetin alfa Hexal AG — HX575 Solution for i.v. injection Containing 1000, 2000 and 4000 IU of rh erythropoietin
  Other Names: Binocrit, Abseamed
  Arms: HX575 epoetin alfa Hexal AG
Drug: ERYPO®, Janssen-Cilag — Solution for i.v. injection
  Other Names: EPREX®; Solution for i.v. injection
  Arms: ERYPO®, Janssen-Cilag

SUMMARY:
This is a double-blind, randomized, multicenter, parallel-group, equivalence study involving about 462 clinically stable hemodialysis patients aged 18 years or above suffering from anemia and treated previously with a stable dose of ERYPO® intravenously.

DETAILED DESCRIPTION:
The primary objective of this Phase III study is the evaluation of therapeutic equivalence of HX575 Hexal AG and a comparator of epoetin alfa, ERYPO® in the maintenance intravenous treatment of renal anemia. Efficacy, dosage and safety of HX575 Hexal AG in the long-term treatment were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Receiving dialysis for at least 6 months (3 times weekly) before screening
* Age: >=18
* Clinically stable, i.e. hemoglobin within the established range (10.0 to 13.0 g/dl) for at least 12 weeks before screening
* Stable intravenous dosage of ERYPO® three times weekly for at least 8 weeks before screening and during screening with a maximal weekly dosage of 300 IU/kg body weight (stable is defined as <25% change (up or down) in weekly dose and no change in frequency over 8 weeks prior screening and 10 weeks prior randomisation)
* Baseline hemoglobin concentration of 10.0 to 13.0 g/dl (mean of two pre-randomization pre-dialysis samples of Hb at visit -2 and visit 1)
* Serum ferritin >=100 µg/l and/or saturated transferrin levels >=20%
* C-reactive protein <15 mg/l (< 5 mg/l: normal; >= 5 mg/l < 10 mg/l: +; >=10mg/l < 100 mg/l: ++; >=100 mg/l: +++)
* Ability to follow study instructions and likely to complete all required visits
* Written informed consent of the patient

Exclusion Criteria:

* Anemia of non-renal causes
* Primary hematologic disorder (e.g. myelodysplastic syndrome, sickle cell anemia, hematological malignancy, hemolytic anemia)
* Evidence of severe hepatic dysfunction (ALT and/or AST above 2 x upper limit of normal range; or gamma-GT above 3 x upper limit of normal range)
* Clinical evidence of current uncontrolled hyperparathyroidism (serum parathyroid hormone >1500 pg/mL).
* Known history of bone marrow disease
* Any red blood cell transfusion(s) during the last 12 weeks before screening or during the screening/baseline period
* Insufficient concomitant iron treatment during the last 2 months before Visit -2
* Uncontrolled hypertension, defined as a predialysis diastolic blood pressure measurement >=110 mmHg during the screening period
* Congestive heart failure [New York Heart Association (NYHA) class III and IV]
* Unstable angina pectoris, active cardiac disease, cardiac infarction during the last six months before screening
* History of blood coagulation disease
* Thrombocytopenia (platelet count <100.000/µl)
* Leukopenia (white blood cell count < 2.000/µl)
* Overt bleeding (acute or chronic bleeding within 2 months of inclusion) or hemolysis
* Evidence of acute infectious disease or serious active inflammatory states within one months before screening (Visit -2) or during the screening/baseline period
* Suspicion or known PRCA (pure red cell aplasia)
* Previously diagnosed HIV or acute hepatitis infection
* Treatment for epilepsy within the past 6 months
* Planned surgery during the next 7 months (except vascular access surgery)
* Any androgen therapy within 2 months before visit -2 and during the study
* Therapy with immunosuppressants or any drug known to affect the hematocrit within 1 month before Visit -2 and during the study
* Clinical evidence of malignant diseases
* Pregnancy, breastfeeding women or women not using adequate birth control measures
* Known history of severe drug related allergies
* Known allergy to one of the ingredients of the test or reference products or hypersensitivity to mammalian-derived products
* Simultaneous participation in another clinical study or participation in a study in the month preceding the start of this study or previously randomized in this study
* Participation in an erythropoietin study in the 3 months preceding screening (visit -2)
* Any other condition which at the investigator´s discretion may put the patient at risk or which may confound the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Haag-Weber, Prof., Principal Investigator — Dialysezentrum Straubing, Germany
Locations (54):
- Austria (9):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Allgemeines Krankenhaus der Barmherzigen Brüder Graz, Graz
  - Dialyseinstitut Graz GmbH, Graz
  - Krankenhaus der Elisabethinen, Graz
  - Universitätsklinik Innsbruck, Klinische Abteilung für Nephrologie, Innsbruck
  - Allgemeines Öffentliches Krankenhaus St. Pölten, I. Med. Abteilung, Sankt Pölten
  - Allgemeines öffentliches Krankenhaus Wiener Neustadt , 2. Interne Abteilung, Vienna
  - Krankenanstalt Rudolfstiftung der Stadt Wien, 3. Med. Abteilung, Vienna
  - Wilhelminenspital der Stadt Wien, Abt. für Nephrologie und Dialyse, Vienna
- Germany (45):
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Aschaffenburg
  - Dialysepraxis Bad Münder, Bad Münder am Deister
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Bad Nauheim
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Bamberg
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Bayreuth
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Bergisch Gladbach
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Berlin
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Bischofswerda
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Bremerhaven
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Coburg
  - Dialysepraxis Drs. Riedasch/Schreiber, Coesfeld
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Deggendorf
  - Dialysepraxis, Donaueschingen
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Eberswalde
  - Dialysepraxis Dr. med. Stefan Holzmann, Erkelenz
  - Dialysepraxis Dr. Möller, Dr. Knee, Essen
  - Dialysepraxis, Freiberg
  - Dialysezentrum, Freiburg im Breisgau
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Fürstenzell
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Greifswald
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Gummersbach
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Günzburg
  - Praxis Dres. Sohn und Schaumann, Hamelin
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Hanover
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Haßfurt
  - Dialysepraxis Dr. med. Stefan Holzmann, Heinsberg
  - Praxis Dr. Kienle, Homberg (Efze)
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Ingolstadt
  - KfH - Prof. Dr. med. Heide Sperschneider, Jena
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Kronach
  - Dialysepraxis Dr. med. Matthias Anders, Leipzig
  - Kfh Kuratorium für Dialyse & Nierentransplantation e.V., 2.Etage, Leipzig
  - KfH Kuratorium für Nierentranplantation und Dialyse e.V., Lohr
  - Dialysepraxis Prof. Rob, Dr. Wilhelm u. Dr. Schümann, Lübeck
  - Dialysepraxis Dr.med. H.-D. Hoffmann, Menden
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, München
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Neuried
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Nördlingen
  - Gemeinschaftspraxis Dr.Steger, Dr.Böhmer, Dr.Kirpal, Nuremberg
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Oberschleißheim
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Plauen
  - Dialysezentrum, Potsdam
  - Praxis Dres.Hartmann, Schiele, Saarbrücken
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Straubing
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Sulzbach-Rosenberg

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 568 patients were screened. 479 were eligible for inclusion and were randomized. 478 patients were started on treatment with either epoetin alfa HX575 Hexal AG or ERYPO®, Janssen-Cilag. As the randomization followed a 2:1 scheme, 314 patients received HX575 Hexal AG and 164 patients received ERYPO®.
Pre-assignment Details: The first part of the study was designed as a double-blind, randomized, multicenter, parallel-group equivalence study and consisted of two phases: Phase I (dose adjustment and maintenance of Hb level; until week 24) followed by Phase II (evaluation period: four week evaluation period to determine the primary efficacy endpoint; weeks 25 until 28).
Groups:
- HX575 Epoetin Alfa Hexal AG: Eligible patients were switched from the comparator to epoetin alfa HX575 Hexal AG in ratio 2:1. Treatment was done intravenously (solution for injection i.v.) in pre-filled syringes for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL. Baseline HB value after 24 weeks was required for efficacy analysis at week 28.
- ERYPO®, Janssen-Cilag: Eligible patients were randomized and continued to be treated intravenously with ERYPO®, Janssen-Cilag in pre-filled syringes (solution for injection i.v.) for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL. Baseline HB value after 24 weeks was required for efficacy analysis at week 28.
Period: Overall Study
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO®, Janssen-Cilag
Started | 314 | 164
Completed | 261 | 142
Not Completed | 53 | 22
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Incl./excl. not fulfilled | 7 | 2
Not completed — Adverse Event | 7 | 6
Not completed — Protocol Violation | 2 | 0
Not completed — Death | 15 | 4
Not completed — Kidney Transplantation (NTX) | 10 | 2
Not completed — Hemoglobulin concentration | 4 | 3
Not completed — Planned operation | 2 | 0
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients who received at least 1 dose of the study medication and for whom at least 1 post-baseline value of the primary endpoint Hb was available. A prerequisite for patients to be included in the Intention To Treat (ITT) population is that they were treated for four weeks with Hb values available during this period.
Groups:
- HX575 Epoetin Alfa Hexal AG: Eligible patients were switched from the comparator to HX575 epoetin alfa Hexal AG in ratio 2:1. Treatment was done intravenously (solution for injection i.v.) in pre-filled syringes for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL. Baseline HB value after 24 weeks was required for efficacy analysis at week 28.
- ERYPO®, Janssen-Cilag: Eligible patients were randomized and continued to be treated with ERYPO® Janssen-Cilag intravenously in pre-filled syringes (solution for injection i.v.) for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL. Baseline HB value after 24 weeks was required for efficacy analysis at week 28.
- Total: Total of all reporting groups
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO®, Janssen-Cilag | Total
Number analyzed (Participants) | 314 | 164 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 145 | 84 | 229
  >=65 years | 169 | 80 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (14.4) | 62.6 (13.8) | 62.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 98 | 236
  Male | 176 | 66 | 242
Region of Enrollment [Number; unit: participants]
  Austria | 70 | 37 | 107
  Germany | 244 | 127 | 371
Body weight [Mean (Standard Deviation); unit: kg] | 76.3 (15.5) | 76.0 (17.7) | 76.2 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Efficacy of HX575 Hexal AG and ERYPO® Janssen-Cilag.
Description: Primary endpoint was the mean absolute change in Hb level between the screening/baseline and the evaluation period. A two-sided 95 % confidence interval for the difference in mean change (mean of evaluation period - mean of screening/baseline period) in Hb between epoetin alfa HX575 Hexal AG and ERYPO® Janssen-Cilag was computed. The difference was estimated from an analysis of a co-variance model including factors treatment, center, mean baseline Hb (<11.5 and ≥11.5 g/dL) as factors and change of the mean weekly dose from screening/baseline to the evaluation period (of HX575 epoetin alfa Hexal AG or ERYPO® Janssen-Cilag) as a covariate. HX575 Hexal AG was considered at least as good as ERYPO® Janssen-Cilag if the 95 % confidence interval of the difference in mean changes in Hb levels between HX575 Hexal AG and ERYPO® Janssen-Cilag lied entirely within the interval [-0.5 g/dL; 0.5 g/dL]. Primary Endpoint was analyzed based on intent-to-treat (ITT) population.
Time Frame: 28 weeks
Population: Primary Endpoint was analyzed based on ITT population: all treated patients with a post baseline hemoglobin value.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Groups:
- ERYPO®, Janssen-Cilag: Eligible patients were randomized and continued to be treated with ERYPO®, Janssen-Cilag in pre-filled syringes intravenously (solution for injection i.v.) for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL. Baseline HB value after 24 weeks was required for efficacy analysis at week 28.
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO®, Janssen-Cilag
Number analyzed (Participants) | 207 | 118
g/dL | 0.147 (0.092) | 0.063 (0.117)
Statistical Analysis 1: Comparison: HX575 Epoetin Alfa Hexal AG; Test type: Equivalence — Therapeutic equivalence was defined as the two-sided 95 % confidence interval of the difference between the two treatment groups lying entirely in the interval -0.5 to 0.5 g/dL. The confidence interval of the difference was calculated based on the least square means (LSMEANS) from an analysis of co-variance model including factors treatment, center, mean baseline Hb level (<11.5 and T11.5 g/dL) as factors and change of the mean weekly dose as a covariate; Point estimate of difference (ANCOVA) = 0.084, 95% CI 2-sided [-0.170 to 0.338]

2. Secondary Outcome: Mean Absolute Change in Hemoglobin Level From the Screening/Baseline Period to the Evaluation Period - ITT Population
Description: The mean absolute change in Hb levels between the screening/baseline period and the evaluation period was analyzed for the intent-to-treat (ITT) population in the same way as the primary efficacy endpoint. A two-sided 95 % confidence interval for the difference in mean change (mean of evaluation period - mean of screening/baseline period) in Hb between HX575 epoetin alfa Hexal AG and ERYPO® Janssen-Cilag was computed. The difference was estimated from an analysis of a co-variance model including factors treatment, center, mean baseline Hb (<11.5 and ≥11.5 g/dL) as factors and change of the mean weekly dose from screening/baseline to the evaluation period (of HX575 epoetin alfa Hexal AG or ERYPO® Janssen-Cilag) as a covariate. HX575 Hexal AG was considered at least as good as ERYPO® Janssen-Cilag if the 95 % confidence interval of the difference in mean changes in Hb levels between HX575 Hexal AG and ERYPO® Janssen-Cilag lied entirely within the interval [-0.5 g/dL; 0.5 g/dL].
Time Frame: 28 weeks
Population: Intent-to-treat population (ITT): all randomized patients who received at least one dose of the study medication and for whom at least one post-baseline value of the primary endpoint Hb was available. A prerequisite to be included in the ITT population was that they were treated for four weeks with Hb values available during this period.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Groups:
- ERYPO®, Janssen-Cilag: Eligible patients were randomized and continued to be treated intravenously with ERYPO® Janssen-Cilag in pre-filled syringes (solution for injection i.v.) for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL. Baseline HB value after 24 weeks was required for efficacy analysis at week 28.
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO®, Janssen-Cilag
Number analyzed (Participants) | 304 | 161
g/dL | 0.003 (0.079) | -0.187 (0.105)
Statistical Analysis 1: Comparison: HX575 Epoetin Alfa Hexal AG vs ERYPO®, Janssen-Cilag; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference LSM of Epo Hexal & Erypo = 0.189, 95% CI 2-sided [-0.039 to 0.418]

ADVERSE EVENTS:
Time Frame: Recording of AEs included periods before first application and until the end of application of study medication. Occurrence of AEs was recorded from time when patient had given his/her informed consent until the final visit of the main study period (visit 28). By definition, AEs starting in the period after first application until the end of the main period were considered to be 'treatment-emergent' AEs. Analysis based on safety population: patients received at least 1 dose of treatment.
Groups:
- HX575 Epoetin Alfa Hexal AG: Eligible patients were switched from the comparator to HX575 epoetin alfa Hexal AG in ratio 2:1 to be intravenously (solution for injection i.v.) treated with HX575 in pre-filled syringes for 24 weeks. The maximum weekly dose was 300 UI/kg body weight (given 1 to 3 times) to maintain hemoglobin levels between 10-13 g/dL. Baseline HB value after 24 weeks was required for efficacy analysis at week 28.
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO®, Janssen-Cilag
All-Cause Mortality (participants affected / at risk) | 19/314 | 5/164
Serious Adverse Events (participants affected / at risk) | 112/314 | 57/164
Other Adverse Events (participants affected / at risk) | 283/314 | 154/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 Epoetin Alfa Hexal AG (N=314) | ERYPO®, Janssen-Cilag (N=164)
Lower respiratory tract and lung infections (Infections and infestations) | 14 (16) | 5 (5)
Bacterial infections NEC (Infections and infestations) | 8 (9) | 1 (1)
Sepsis, bacteraemia and viraemia (Infections and infestations) | 7 (8) | 1 (1)
Infections NEC (Infections and infestations) | 4 (4) | 2 (2)
Abdominal and gastrointestinal infections (Infections and infestations) | 4 (6) | 0 (0)
Bone and joint infections (Infections and infestations) | 2 (2) | 1 (1)
Streptococcal infections (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infections (Infections and infestations) | 2 (3) | 0 (0)
Cardiac infections (Infections and infestations) | 1 (1) | 0 (0)
Influenza viral infections (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal infections (Infections and infestations) | 1 (1) | 0 (0)
Skin structures and soft tissue infections (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infections (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infections (Infections and infestations) | 0 (0) | 1 (1)
Vascular infections (Infections and infestations) | 1 (1) | 0 (0)
Viral infections NEC (Infections and infestations) | 1 (1) | 0 (0)
Cardiac and vascular procedural complications (Injury, poisoning and procedural complications) | 24 (27) | 14 (18)
Lower limb fractures and dislocations (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cerebral injuries NEC (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fractures and dislocations NEC (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injuries NEC (incl traumatic amputation) (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Device failure and malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device related complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Site specific injuries NEC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic cage fractures and dislocations (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fractures and dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ischaemic coronary artery disorders (Cardiac disorders) | 17 (24) | 7 (8)
Rate and rhythm disorders NEC (Cardiac disorders) | 6 (6) | 3 (3)
Heart failures NEC (Cardiac disorders) | 4 (6) | 1 (1)
Supraventricular arrhythmias (Cardiac disorders) | 5 (6) | 0 (0)
Ventricular arrhythmias and cardiac arrest (Cardiac disorders) | 4 (4) | 0 (0)
Coronary artery disorders NEC (Cardiac disorders) | 1 (1) | 2 (2)
Aortic valvular disorders (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorders NEC (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomyopathies (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral vasoconstriction, necrosis and vascular insufficiency (Vascular disorders) | 8 (8) | 2 (2)
Accelerated and malignant hypertension (Vascular disorders) | 5 (5) | 1 (1)
Aneurysms and dissections non-site specific (Vascular disorders) | 1 (1) | 2 (2)
Non-site specific necrosis and vascular insufficiency NEC (Vascular disorders) | 2 (2) | 1 (1)
Vascular hypertensive disorders NEC (Vascular disorders) | 2 (2) | 1 (1)
Vascular hypotensive disorders (Vascular disorders) | 2 (2) | 1 (1)
Peripheral embolism and thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haemorrhages NEC (Vascular disorders) | 0 (0) | 1 (1)
Site specific necrosis and vascular insufficiency NEC (Vascular disorders) | 1 (1) | 0 (0)
Vena caval embolism and thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Acute and chronic pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcers and perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (excl infective) (Gastrointestinal disorders) | 1 (1) | 2 (2)
Non-site specific gastrointestinal haemorrhages (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diverticula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal inflammatory disorders NEC (Gastrointestinal disorders) | 1 (1) | 1 (1)
Benign neoplasms gastrointestinal (excl oral cavity) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcers and perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspeptic signs and symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal signs and symptoms NEC (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal spastic and hypermotility disorders (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal vascular occlusion and infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids and gastrointestinal varices (excl oesophageal) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernias (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ulcers and perforation NEC (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal and retroperitoneal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal and retroperitoneal haemorrhages (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchospasm and obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pulmonary oedemas (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lower respiratory tract inflammatory and immunologic conditions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failures (excl neonatal) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal disorders NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Parenchymal lung disorders NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary thrombotic and embolic conditions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Central nervous system haemorrhages and cerebrovascular accidents (Nervous system disorders) | 5 (5) | 2 (2)
Central nervous system vascular disorders NEC (Nervous system disorders) | 3 (3) | 0 (0)
Seizures and seizure disorders NEC (Nervous system disorders) | 0 (0) | 2 (2)
Coma states (Nervous system disorders) | 1 (1) | 0 (0)
Disturbances in consciousness NEC (Nervous system disorders) | 1 (1) | 0 (0)
Mononeuropathies (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis and paresis (excl congenital and cranial nerve) (Nervous system disorders) | 0 (0) | 1 (1)
Febrile disorders (General disorders) | 1 (1) | 1 (1) — General disorders and administrative site conditions
Implant and catheter site reactions (General disorders) | 1 (1) | 1 (1) — General disorders and administration site conditions
Body temperature perception (General disorders) | 0 (0) | 1 (1) — General disorders and administration site conditions
Death and sudden death (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
General signs and symptoms NEC (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Healing abnormal NEC (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Trophic disorders (General disorders) | 0 (0) | 1 (1) — General disorders and administration site conditions
Colonic neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to specified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory tract small cell carcinomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin neoplasms malignant and unspecified (excl melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft tissue neoplasms benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 3 (4) | 3 (3)
Cholestasis and jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthropathies NEC (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathies (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue ulcerations (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dermal and epidermal conditions NEC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal disorders NEC (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder infections and inflammations (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal obstructive disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal vascular and ischaemic conditions (Renal and urinary disorders) | 0 (0) | 1 (1)
Arterial therapeutic procedures (excl aortic) (Surgical and medical procedures) | 1 (1) | 1 (1)
Vascular therapeutic procedures NEC (Surgical and medical procedures) | 2 (2) | 0 (0)
Joint therapeutic procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypoglycaemic conditions NEC (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Calcium metabolism disorders NEC (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (incl subtypes) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Total fluid volume increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Carbohydrate tolerance analyses (incl diabetes) (Investigations) | 1 (1) | 0 (0)
ECG investigations (Investigations) | 1 (1) | 0 (0)
Gastrointestinal histopathology procedures (Investigations) | 1 (1) | 0 (0)
Hyperparathyroid disorders (Endocrine disorders) | 2 (2) | 0 (0)
Confusion and disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Depressive disorders (Psychiatric disorders) | 1 (1) | 0 (0)
Anaemias NEC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Inner ear signs and symptoms (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataracts (excl congenital) (Eye disorders) | 1 (1) | 0 (0)
Transplant rejections (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 Epoetin Alfa Hexal AG (N=314) | ERYPO®, Janssen-Cilag (N=164)
Nasopharyngitis (Infections and infestations) | 55 (73) | 35 (41)
Bronchitis (Infections and infestations) | 28 (34) | 19 (20)
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 49 (224) | 23 (100)
Procedural hypotension (Injury, poisoning and procedural complications) | 44 (137) | 23 (60)
Procedural hypertension (Injury, poisoning and procedural complications) | 16 (76) | 10 (39)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 18 (20) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 63 (85) | 22 (23)
Vomiting (Gastrointestinal disorders) | 27 (36) | 18 (21)
Nausea (Gastrointestinal disorders) | 30 (43) | 14 (20)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 77 (276) | 38 (86)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (19) | 11 (16)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 11 (14)
Hypotension (Vascular disorders) | 48 (142) | 20 (26)
Hypertension (Vascular disorders) | 29 (62) | 9 (17)
Headache (Nervous system disorders) | 29 (53) | 13 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 14 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (20) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes